CLINICAL TRIAL: NCT01556178
Title: Collection of Blood and Cerebrospinal Fluid for Pediatric Brain Tumor Research
Brief Title: Blood and Cerebrospinal Fluid for Pediatric Brain Tumor Research
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Rishi Lulla, Principal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2011-14612
Record Dates: First submitted 2012-02-24; First posted 2012-03-16 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Hydrocephalus
Keywords: Hydrocephalus; Survivin; miRNA
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood and cerebrospinal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children without central nervous system tumors: Children without central nervous system tumors between the ages of 1 year and 21 years who are undergoing a neurosurgical procedure to address hydrocephalus

SUMMARY:
In normal patients, blood and cerebrospinal fluid (CSF) contain circulating cells and other molecules such as proteins and nucleic acids. In patients with central nervous system (CNS) and other conditions, the levels of these molecules may be altered. In several other studies at our institution, the investigators are investigating such molecules in tumor specimens as well as the blood and cerebrospinal fluid of pediatric patients with CNS tumors. However, these levels are difficult to interpret without comparing them to levels in patients without CNS tumors. The investigators propose a study to collect small amounts of blood and cerebrospinal fluid from pediatric patients without CNS tumors who are undergoing a diagnostic or therapeutic neurosurgical procedure aimed at addressing altered CSF dynamics.

ELIGIBILITY:
Inclusion Criteria:

* Children without central nervous system tumors who are undergoing a neurosurgical procedure to address hydrocephalus during which CSF will be obtained
* Between the ages of 1 year and 21 years
* Patients must be having blood draws, lumbar punctures or CSF sampling from Ommaya reservoirs or VPS as part of routine clinical care.

Exclusion Criteria:

* Patients who do not require routine blood draws and/or CSF collection as part of their routine clinical care
* Patients who are considered too ill to participate as determined by their treating physician
* Patients with documented bacterial of viral infections of the CSF, brain parenchyma and/or neurosurgical devices and/or
* Patients with suspected de-myelinating conditions
* Patients who are pregnant or lactating.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children without central nervous system tumors between the ages of 1 year and 21 years who are undergoing a neurosurgical procedure to address hydrocephalus during which CSF will be obtained will be considered
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
levels of miRNAs in the blood and CSF | 2 yrs

SECONDARY OUTCOMES:
Survivin and biologic markers levels in the CSF and blood | 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Lulla, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Fernandez-L A, Northcott PA, Taylor MD, Kenney AM. Normal and oncogenic roles for microRNAs in the developing brain. Cell Cycle. 2009 Dec 15;8(24):4049-54. doi: 10.4161/cc.8.24.10243. Epub 2009 Dec 5. PMID 19901543
- [Background] Mitchell PS, Parkin RK, Kroh EM, Fritz BR, Wyman SK, Pogosova-Agadjanyan EL, Peterson A, Noteboom J, O'Briant KC, Allen A, Lin DW, Urban N, Drescher CW, Knudsen BS, Stirewalt DL, Gentleman R, Vessella RL, Nelson PS, Martin DB, Tewari M. Circulating microRNAs as stable blood-based markers for cancer detection. Proc Natl Acad Sci U S A. 2008 Jul 29;105(30):10513-8. doi: 10.1073/pnas.0804549105. Epub 2008 Jul 28. PMID 18663219
- [Background] Taylor DD, Gercel-Taylor C. MicroRNA signatures of tumor-derived exosomes as diagnostic biomarkers of ovarian cancer. Gynecol Oncol. 2008 Jul;110(1):13-21. doi: 10.1016/j.ygyno.2008.04.033. PMID 18589210
- [Background] Lawrie CH, Gal S, Dunlop HM, Pushkaran B, Liggins AP, Pulford K, Banham AH, Pezzella F, Boultwood J, Wainscoat JS, Hatton CS, Harris AL. Detection of elevated levels of tumour-associated microRNAs in serum of patients with diffuse large B-cell lymphoma. Br J Haematol. 2008 May;141(5):672-5. doi: 10.1111/j.1365-2141.2008.07077.x. Epub 2008 Mar 3. PMID 18318758
- [Background] Huang Z, Huang D, Ni S, Peng Z, Sheng W, Du X. Plasma microRNAs are promising novel biomarkers for early detection of colorectal cancer. Int J Cancer. 2010 Jul 1;127(1):118-26. doi: 10.1002/ijc.25007. PMID 19876917
- [Background] Ng EK, Chong WW, Jin H, Lam EK, Shin VY, Yu J, Poon TC, Ng SS, Sung JJ. Differential expression of microRNAs in plasma of patients with colorectal cancer: a potential marker for colorectal cancer screening. Gut. 2009 Oct;58(10):1375-81. doi: 10.1136/gut.2008.167817. Epub 2009 Feb 6. PMID 19201770
- [Background] Heneghan HM, Miller N, Lowery AJ, Sweeney KJ, Kerin MJ. MicroRNAs as Novel Biomarkers for Breast Cancer. J Oncol. 2009;2009:950201. doi: 10.1155/2010/950201. Epub 2009 Jul 20. PMID 19639033
- [Background] Zhu W, Qin W, Atasoy U, Sauter ER. Circulating microRNAs in breast cancer and healthy subjects. BMC Res Notes. 2009 May 19;2:89. doi: 10.1186/1756-0500-2-89. PMID 19454029
- [Background] Chakravarti A, Noll E, Black PM, Finkelstein DF, Finkelstein DM, Dyson NJ, Loeffler JS. Quantitatively determined survivin expression levels are of prognostic value in human gliomas. J Clin Oncol. 2002 Feb 15;20(4):1063-8. doi: 10.1200/JCO.2002.20.4.1063. PMID 11844831
- [Background] Fangusaro JR, Jiang Y, Holloway MP, Caldas H, Singh V, Boue DR, Hayes J, Altura RA. Survivin, Survivin-2B, and Survivin-deItaEx3 expression in medulloblastoma: biologic markers of tumour morphology and clinical outcome. Br J Cancer. 2005 Jan 31;92(2):359-65. doi: 10.1038/sj.bjc.6602317. PMID 15655550
- [Background] Ikeguchi M, Kaibara N. survivin messenger RNA expression is a good prognostic biomarker for oesophageal carcinoma. Br J Cancer. 2002 Oct 7;87(8):883-7. doi: 10.1038/sj.bjc.6600546. PMID 12373603
- [Background] Ikeguchi M, Ueda T, Sakatani T, Hirooka Y, Kaibara N. Expression of survivin messenger RNA correlates with poor prognosis in patients with hepatocellular carcinoma. Diagn Mol Pathol. 2002 Mar;11(1):33-40. doi: 10.1097/00019606-200203000-00007. PMID 11854600
- [Background] Monzo M, Rosell R, Felip E, Astudillo J, Sanchez JJ, Maestre J, Martin C, Font A, Barnadas A, Abad A. A novel anti-apoptosis gene: Re-expression of survivin messenger RNA as a prognosis marker in non-small-cell lung cancers. J Clin Oncol. 1999 Jul;17(7):2100-4. doi: 10.1200/JCO.1999.17.7.2100. PMID 10561264
- [Background] Mori A, Wada H, Nishimura Y, Okamoto T, Takemoto Y, Kakishita E. Expression of the antiapoptosis gene survivin in human leukemia. Int J Hematol. 2002 Feb;75(2):161-5. doi: 10.1007/BF02982021. PMID 11939262
- [Background] Sarela AI, Verbeke CS, Ramsdale J, Davies CL, Markham AF, Guillou PJ. Expression of survivin, a novel inhibitor of apoptosis and cell cycle regulatory protein, in pancreatic adenocarcinoma. Br J Cancer. 2002 Mar 18;86(6):886-92. doi: 10.1038/sj.bjc.6600133. PMID 11953819
- [Background] Takamizawa S, Scott D, Wen J, Grundy P, Bishop W, Kimura K, Sandler A. The survivin:fas ratio in pediatric renal tumors. J Pediatr Surg. 2001 Jan;36(1):37-42. doi: 10.1053/jpsu.2001.20000. PMID 11150435
- [Background] Adida C, Berrebi D, Peuchmaur M, Reyes-Mugica M, Altieri DC. Anti-apoptosis gene, survivin, and prognosis of neuroblastoma. Lancet. 1998 Mar 21;351(9106):882-3. doi: 10.1016/S0140-6736(05)70294-4. No abstract available. PMID 9525374
- [Background] Islam A, Kageyama H, Takada N, Kawamoto T, Takayasu H, Isogai E, Ohira M, Hashizume K, Kobayashi H, Kaneko Y, Nakagawara A. High expression of Survivin, mapped to 17q25, is significantly associated with poor prognostic factors and promotes cell survival in human neuroblastoma. Oncogene. 2000 Feb 3;19(5):617-23. doi: 10.1038/sj.onc.1203358. PMID 10698506
- [Background] Ito R, Asami S, Motohashi S, Ootsuka S, Yamaguchi Y, Chin M, Shichino H, Yoshida Y, Nemoto N, Mugishima H, Suzuki T. Significance of survivin mRNA expression in prognosis of neuroblastoma. Biol Pharm Bull. 2005 Apr;28(4):565-8. doi: 10.1248/bpb.28.565. PMID 15802787